CLINICAL TRIAL: NCT05779059
Title: Prasugrel Or Ticagrelor De-escalation in Non-ST-elevation Acute Coronary Syndrome
Brief Title: Prasugrel Or Ticagrelor De-escalation in NSTE-ACS
Acronym: PROTEUS
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Collegium Medicum w Bydgoszczy (Other)
Responsible Party: Principal Investigator, Piotr Adamski, MD, PhD, Associate Professor, Collegium Medicum w Bydgoszczy
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2023/01
Record Dates: First submitted 2023-03-09; First posted 2023-03-22 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2023-03

CONDITIONS: Non ST Segment Elevation Acute Coronary Syndrome; Non-ST-Segment Elevation Myocardial Infarction (NSTEMI); Unstable Angina
Keywords: acute coronary syndrome; de-escalation; prasugrel; ticagrelor
MeSH Terms: conditions — Non-ST Elevated Myocardial Infarction; Angina, Unstable; Acute Coronary Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Initial ticagrelor (Experimental): All patients will receive standard 180 mg loading dose of ticagrelor, followed by a standard maintenance dose of 90 mg bid for 30 days, after which de-escalation to 60 mg bid will take place and this dosing will be maintained for 15 days. At day 45 all patients will be loaded with standard 60 mg dose of prasugrel followed by reduced maintenance dose of 5 mg qd for 15 days. At day 60 all patients will be switched back to guideline recommended antiplatelet therapy.
  Interventions: Drug: De-escalation to ticagrelor 60 mg at day 30; Drug: Switch to prasugrel 5 mg at day 45
- Initial prasugrel (Experimental): All patients will receive standard 60 mg loading dose of prasugrel, followed by a standard maintenance dose 10 mg qd for 30 days, after which de-escalation to 5 mg qd will take place and this dosing will be maintained for 15 days. At day 45 patients will be loaded with standard 180 mg dose of ticagrelor followed by reduced maintenance dose of 60 mg bid for 15 days. At day 60 all patients will be switched back to guideline recommended antiplatelet therapy.
  Interventions: Drug: De-escalation to prasugrel 5 mg at day 30; Drug: Switch to ticagrelor 60 mg at day 45

INTERVENTIONS:
Drug: De-escalation to ticagrelor 60 mg at day 30 — Change of P2Y12 receptor antagonist regimen to ticagrelor 60 mg bid at day 30.
  Arms: Initial ticagrelor
Drug: De-escalation to prasugrel 5 mg at day 30 — Change of P2Y12 receptor antagonist regimen to prasugrel 5 mg qd at day 30.
  Arms: Initial prasugrel
Drug: Switch to ticagrelor 60 mg at day 45 — Switch to ticagrelor 60 mg bid at day 45.
  Arms: Initial prasugrel
Drug: Switch to prasugrel 5 mg at day 45 — Switch to prasugrel 5 mg qd at day 45.
  Arms: Initial ticagrelor

SUMMARY:
The PROTEUS study is a randomized, cross-over, open-label, pharmacodynamic trial designed to compare the antiplatelet effect of reduced maintenance doses of prasugrel and ticagrelor in stable patients who recently had non-ST-elevation acute coronary syndrome (non-ST-elevation myocardial infarction or unstable angina).

ELIGIBILITY:
Inclusion Criteria:

* provision of informed consent prior to any study specific procedures
* diagnosis of non-ST-segment elevation acute coronary syndrome (non-ST-segment elevation myocardial treatment or unstable angina)
* male or non-pregnant female, aged 18-75 years old

Exclusion Criteria:

* known hypersensitivity to ticagrelor or prasugrel
* presence of contraindications for ticagrelor or prasugrel
* current treatment with oral anticoagulant or chronic therapy with low-molecular-weight heparin
* history of ischemic stroke or transient ischemic attack
* history of intracranial hemorrhage
* recent gastrointestinal bleeding (within 30 days)
* history of moderate or severe hepatic impairment
* history of major surgery or severe trauma (within 3 months)
* patient required dialysis
* concomitant therapy with strong CYP3A inhibitors (ketoconazole, itraconazole, voriconazole, telithromycin, clarithromycin, nefazadone, ritonavir, saquinavir, nelfinavir, indinavir, atazanavir) or strong CYP3A inducers (rifampicin, phenytoin, carbamazepine, dexamethasone, phenobarbital) within 14 days and during study treatment
* body weight below 60 kg

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-04-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Platelet Reactivity Assessed with Multiple Electrode Aggregometry | day 15 of using reduced maintenance dose of prasugrel or ticagrelor
  Platelet Reactivity Assessed with Multiple Electrode Aggregometry will be evaluated after 15 days of using reduced maintenance dose of prasugrel or ticagrelor.

SECONDARY OUTCOMES:
Platelet Reactivity Assessed with the VerifyNow assay | day 15 of using reduced maintenance dose of prasugrel or ticagrelor
  Platelet Reactivity Assessed with the VerifyNow assay will be evaluated after 15 days of using reduced maintenance dose of prasugrel or ticagrelor.
High Platelet Reactivity according to Multiple Electrode Aggregometry | day 15 of using reduced maintenance dose of prasugrel or ticagrelor
  Percentage of Patients With High Platelet Reactivity according to Multiple Electrode Aggregometry after 15 days of using reduced maintenance dose of prasugrel or ticagrelor.
High Platelet Reactivity according to the VerifyNow assay | day 15 of using reduced maintenance dose of prasugrel or ticagrelor
  Percentage of Patients With High Platelet Reactivity according to the VerifyNow assay after 15 days of using reduced maintenance dose of prasugrel or ticagrelor.

CONTACTS AND LOCATIONS:
Overall Officials: Piotr Adamski, MD, PhD, Principal Investigator — CM UMK
Locations (1):
- Department of Cardiology, Dr. A. Jurasz University Hospital, Collegium Medicum, Nicolaus Copernicus University, Bydgoszcz, Kuyavian-Pomeranian Voivodeship, Poland